CLINICAL TRIAL: NCT03622385
Title: Exploration of DNA Methylation as a Marker for Early Detection of High Grade Serous Epithelial Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 018-530
Record Dates: First submitted 2018-07-30; First posted 2018-08-09 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Epithelial Ovarian Cancer
Keywords: DNA Methylation; DNA Biomarkers; Pelvic Mass
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — DNA Methylation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — During the retrospective phase of the study, archival tissue samples will undergo genome-scale DNA methylation analysis (Reduced Representation Bisulfite Sequencing, RRBS).
  Blood and tissue samples will be obtained from patients who consent to enroll in the prospective phase of this study. Samples will undergo a biomarker validation by performing quantitative RT-PCRs for methylated DNA biomarkers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients diagnosed with Serous Epithelial Ovarian Cancer: Discovery Cohort: patients who were diagnosed with serous epithelial ovarian cancer whose tissue specimens were previously collected.
  Validation Cohort: patients who are scheduled for a diagnostic laparoscopic biopsy for an undiagnosed pelvic mass that is determined to be cancerous.
  Interventions: Other: DNA Methylation
- Normal patients: Discovery Cohort: patients who were determined to have normal ovarian tissue specimens that were previously collected.
  Validation Cohort: patients who are scheduled for a diagnostic laparoscopic biopsy for an undiagnosed pelvic mass that is determined to not be cancerous.
  Interventions: Other: DNA Methylation

INTERVENTIONS:
Other: DNA Methylation — No intervention will be performed. Blood and tissue samples will be analyzed for biomarkers that may be used to develop a diagnostic panel for early detection and diagnosis of high grade serous epithelial ovarian cancer.

SUMMARY:
The purpose of this study is to determine if there are markers in plasma that can be used to develop a diagnostic panel for early detection and diagnosis of high grade serous epithelial ovarian cancer.

DETAILED DESCRIPTION:
This study has two phases: "Discovery" cohort and "Validation" cohort.

The "Discovery" phase of this study will obtain tissue samples in a retrospective manner. The investigators will perform genome-scale DNA Methylation analysis to obtain a panel of candidate methylated DNA biomarkers. Twenty archival primary serous epithelial ovarian cancer and twenty archival normal ovarian and salpingeal tissues will be identified by running a report of diagnosis.

During the "Validation" phase of this study, blood and tissue samples will be obtained in a prospective manner. The patients will be undergoing consultation for undiagnosed pelvic mass and are being scheduled for a diagnostic laparoscopic biopsy. At the time of their consultation, patients will be recruited and consented for this phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years of age and older
* Women with an undiagnosed pelvic mass who need to undergo diagnostic laparoscopic surgery

Exclusion Criteria:

* Male
* Under 18 years of age
* Women who can not give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The investigators are studying biomarkers for the early detection of ovarian cancer. Patients will need to have had ovaries.
Study Population: Patients who will be recruited for the prospective phase of the study will be women, 18 years of age or older, who have an undiagnosed pelvic mass who need to undergo diagnostic laparoscopic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
Identification of DNA markers using HiSeq Genome Analyzer that can predict Serous Epithelial Ovarian Cancer | 2 years
  Isolate DNA using QiaAMp DNA mini kits from tissue and plasma samples from subjects with serous epithelial ovarian cancer and normal subjects and then sequence the DNA using HiSeq Genome Analyzer. The investigators will identify the sequence reads using Illumina base-calling software and analyze them using Zymo Research proprietary analysis pipeline to identify differences in genomic expression in normal subjects compared to subjects with Serous Epithelial Ovarian Cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Jack Stecher, MD, Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cancer Genome Atlas Network. Comprehensive molecular portraits of human breast tumours. Nature. 2012 Oct 4;490(7418):61-70. doi: 10.1038/nature11412. Epub 2012 Sep 23. PMID 23000897
- [Background] Lu KH. Screening for Ovarian Cancer in Asymptomatic Women. JAMA. 2018 Feb 13;319(6):557-558. doi: 10.1001/jama.2017.21894. No abstract available. PMID 29450509
- [Background] Melnikov A, Scholtens D, Godwin A, Levenson V. Differential methylation profile of ovarian cancer in tissues and plasma. J Mol Diagn. 2009 Jan;11(1):60-65. doi: 10.2353/jmoldx.2009.080072. Epub 2008 Dec 12. PMID 19074590
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2018. CA Cancer J Clin. 2018 Jan;68(1):7-30. doi: 10.3322/caac.21442. Epub 2018 Jan 4. PMID 29313949
- [Background] Warton K, Samimi G. Methylation of cell-free circulating DNA in the diagnosis of cancer. Front Mol Biosci. 2015 Apr 22;2:13. doi: 10.3389/fmolb.2015.00013. eCollection 2015. PMID 25988180
- [Result] Buys SS, Partridge E, Greene MH, Prorok PC, Reding D, Riley TL, Hartge P, Fagerstrom RM, Ragard LR, Chia D, Izmirlian G, Fouad M, Johnson CC, Gohagan JK; PLCO Project Team. Ovarian cancer screening in the Prostate, Lung, Colorectal and Ovarian (PLCO) cancer screening trial: findings from the initial screen of a randomized trial. Am J Obstet Gynecol. 2005 Nov;193(5):1630-9. doi: 10.1016/j.ajog.2005.05.005. PMID 16260202
- [Result] Jacobs IJ, Menon U, Ryan A, Gentry-Maharaj A, Burnell M, Kalsi JK, Amso NN, Apostolidou S, Benjamin E, Cruickshank D, Crump DN, Davies SK, Dawnay A, Dobbs S, Fletcher G, Ford J, Godfrey K, Gunu R, Habib M, Hallett R, Herod J, Jenkins H, Karpinskyj C, Leeson S, Lewis SJ, Liston WR, Lopes A, Mould T, Murdoch J, Oram D, Rabideau DJ, Reynolds K, Scott I, Seif MW, Sharma A, Singh N, Taylor J, Warburton F, Widschwendter M, Williamson K, Woolas R, Fallowfield L, McGuire AJ, Campbell S, Parmar M, Skates SJ. Ovarian cancer screening and mortality in the UK Collaborative Trial of Ovarian Cancer Screening (UKCTOCS): a randomised controlled trial. Lancet. 2016 Mar 5;387(10022):945-956. doi: 10.1016/S0140-6736(15)01224-6. Epub 2015 Dec 17. PMID 26707054
- [Result] Liggett TE, Melnikov A, Yi Q, Replogle C, Hu W, Rotmensch J, Kamat A, Sood AK, Levenson V. Distinctive DNA methylation patterns of cell-free plasma DNA in women with malignant ovarian tumors. Gynecol Oncol. 2011 Jan;120(1):113-20. doi: 10.1016/j.ygyno.2010.09.019. Epub 2010 Nov 6. PMID 21056906
- [Result] Survival Rates for Ovarian Cancer by Stage. American Cancer society Website, February 2, 2016. https://www.cancer.org/cancer/ovarian-cancer/detection-diagnosis-staging/survival-rates.html